CLINICAL TRIAL: NCT01722591
Title: A Prospective, Multicenter, Uncontrolled Study to Evaluate the Safety and Efficacy of the Cardiapex Percutaneous Trans-apical Access and Closure System
Brief Title: Safety and Efficacy Study of the Cardiapex Percutaneous Trans-apical Access and Closure System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiapex Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CLN-PRO-01
Record Dates: First submitted 2012-11-02; First posted 2012-11-07 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Transapical Transcatheter Aortic Valve Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiapex device (Experimental): Use of the Cardiapex device in the context of transapical TAVI procedures
  Interventions: Device: Cardiapex device

INTERVENTIONS:
Device: Cardiapex device — Cardiapex percutaneous transapical access and closure system

SUMMARY:
A prospective, multicenter, uncontrolled study to evaluate the safety and efficacy of the Cardiapex percutaneous trans-apical access and closure system. The Cardiapex device intended for percutaneous access and closure of the left ventricular apex in conjunction with transapical Transcatheter Aortic Valve Implantation (TAVI).

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for transapical TAVI
* Patient ≥ 70 years of age
* Patient able to give informed written consent
* Patient able to attend follow up examinations

Exclusion Criteria:

* Scheduled concomitant non-TAVI cardiac procedure
* Patient with Left Ventricular Ejection Fraction (LVEF) < 30% at time of enrollment
* Patient with known apical infarcted area
* Patient with a distinct large vessel right at the anatomical apex9 (based on pre-operative coronary angiography
* Patients with known lung tissue surrounding the apex and possibly interfering with the in-out puncture (based on preoperative gated CT assessment
* Patient with contra-indications to transapical TAVI
* Patient's inability to tolerate or comply with normal post-surgical drug regimen
* Patient's inability to comply with required follow-ups, including echocardiography
* Patient participation in other clinical trials within previous month

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Successful performance of percutaneous transapical TAVI defined as: "Successful percutaneous transapical access and deployment of a single prosthetic heart valve" | Outcome measure assessed during the TAVI surgical procedure - an average of 3 hours

SECONDARY OUTCOMES:
≤30 day apical bleeding requiring surgical intervention | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Kerckhoff Clinic, Bad Nauheim
  - Hamburg University Heart Center, Hamburg